CLINICAL TRIAL: NCT03003819
Title: A Prospective, Randomized, Controlled, Multi-center Evaluation of Extraction Socket Management Comparing Two Socket Sealing Collagen Matrices
Brief Title: A Comparison of Two Socket Sealing Collagen Matrices for Extraction Socket Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGuire Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPNA0001-2016
Record Dates: First submitted 2016-12-18; First posted 2016-12-28 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Collagen Wound Dressing (Active Comparator): Bovine collagen sponge used to control bleeding, stabilize blood clots and protect dental wounds
  Interventions: Device: Control Collagen Wound Dressing
- Test Collagen Matrix (Active Comparator): Bilayer, porcine collagen matrix for soft tissue regeneration used as a socket seal in extraction socket grafting
  Interventions: Device: Test Collagen Matrix

INTERVENTIONS:
Device: Control Collagen Wound Dressing — Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic and local anesthetic, minimally traumatic extraction will be performed with periotomes . After degranulation and bone graft placement, control or test biomaterial will be placed according to the randomization schedule and surgical instructions for each biomaterial.
  Arms: Control Collagen Wound Dressing
Device: Test Collagen Matrix — Following resolution of any periodontal issues in the region of study and administration of pre-surgical antibiotic and local anesthetic, minimally traumatic extraction will be performed with periotomes . After degranulation and bone graft placement, control or test biomaterial will be placed according to the randomization schedule and surgical instructions for each biomaterial.
  Arms: Test Collagen Matrix

SUMMARY:
A prospective RCT of intact extractions with delayed implant placement comparing extraction socket management effectiveness and office economics of two collagen matrices. Soft tissue wound healing will be assessed out to 4-months post-operative, when implants will be placed.

DETAILED DESCRIPTION:
A prospective, randomized, multi-center, controlled clinical study of intact extractions (bony dehiscences <1/3 socket apico-coronal and mesial-distal dimension) with delayed implant placement. Study objective: to compare extraction socket management effectiveness and office economics of a frequently used wound dressing (control) with a soft tissue augmentation matrix (test) in 32-64 subjects 18 -75 years of age with intact (bony dehiscence, if present, < 1/3 socket dimension) extractions intended for dental implant replacement. Following screening subjects will undergo tooth extraction and randomization to either the control or test therapy. After treatment, subjects will be followed until 4- months, the time of implant placement. Primary outcome: soft tissue wound healing measured by (1) gap closure and (2) graft containment at all time points.

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated for anterior tooth extraction (from premolars forward) intended for implant placement.
* Subjects with essentially intact extraction sockets - bony dehiscences < 1/3 the depth of socket and mesial-distal width of tooth socket
* Subjects will have read, understood and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
* Subjects must be able and willing to follow study procedures and instructions

Exclusion Criteria:

* Subjects with healing disorders (i.e., diabetes mellitus, cancer, HIV, bone metabolic diseases) that could compromise wound healing and/ or preclude implant surgery; or who are currently receiving or have received within two months prior to study entry, systemic corticosteroids, immunosuppressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery.
* Subjects taking intramuscular or intravenous bisphosphonates.
* Subjects who have a known allergy or sensitivity to collagen.
* Subjects with acute, suppurative lesions with pain, swelling and apical lesions > 5mm will be excluded, though antibiotic prophylaxis may be employed to reduce infection and provide possible subject reconsideration for inclusion.
* Heavy smokers/tobacco users defined as those smoking ≥ 10 cigarettes or ≥ 4 cigars or ≥ 4 pipes per day. For non-heavy smokers, smoking ≥ 10 cigarettes or ≥ 4 cigars or ≥ 4 pipes per day is prohibited for the duration of the study.
* Female subjects who are pregnant or lactating, or who intend to become pregnant during the study duration
* Subjects participating in other clinical studies involving therapeutic intervention (either medical or dental).
* Subjects, who in the opinion of the Investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Socket Soft Tissue Gap Closure - linear measures buccal-lingual in millimeters | 4-months
  Longitudinal extraction socket soft tissue gap closure measured buccal-lingual from baseline to 4-months.

SECONDARY OUTCOMES:
Socket Soft Tissue Gap Closure - linear measures mesial-distal | 4-months
  Longitudinal extraction socket soft tissue gap closure measured mesial-distal from baseline to 4-months.
Graft Containment as observed by subject and examiner (yes/ no) | 4-months
Inflammation Score (Loe and Sillness) | 4-months
Biomaterial Integrity - 4-point scale | 4-months
  Score 0-4, 0 = biomaterial completely present, 4 = no evidence of biomaterial/ complete granulation or other tissue
Tissue Thickness - probe show-thru at baseline and biopsy measure in millimeters at 4-months | 4-months
  Soft tissue thickness is measured using probe "show-thru" (tissue transparency) at baseline and soft tissue biopsy at the implant site immediately prior to implant placement

CONTACTS AND LOCATIONS:
Overall Officials: Todd V Scantlebury, BS, Study Director — The McGuire Institute
Locations (1):
- Seven Lakes Periodontics, Fenton, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thoma DS, Sancho-Puchades M, Ettlin DA, Hammerle CH, Jung RE. Impact of a collagen matrix on early healing, aesthetics and patient morbidity in oral mucosal wounds - a randomized study in humans. J Clin Periodontol. 2012 Feb;39(2):157-65. doi: 10.1111/j.1600-051X.2011.01823.x. Epub 2011 Dec 6. PMID 22145767
- [Background] Sclar AG. Strategies for management of single-tooth extraction sites in aesthetic implant therapy. J Oral Maxillofac Surg. 2004 Sep;62(9 Suppl 2):90-105. doi: 10.1016/j.joms.2004.06.041. PMID 15332186